CLINICAL TRIAL: NCT01391143
Title: A Phase 1 Dose Escalation Study of MGA271 in Refractory Cancer
Brief Title: Safety Study of MGA271 in Refractory Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGA271-01
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer; Melanoma; Renal Cell Carcinoma; Triple-negative Breast Cancer; Head and Neck Cancer; Bladder Cancer; Non-small Cell Lung Cancer
Keywords: Prostate cancer; Melanoma; Renal cell carcinoma; Triple-negative breast cancer; Head and neck cancer; Bladder cancer; Non-small cell lung cancer; Squamous cell carcinoma
MeSH Terms: conditions — Prostatic Neoplasms; Melanoma; Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Head and Neck Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MGA271 (Experimental): Fc-optimized, humanized monoclonal antibody
  Interventions: Biological: MGA271

INTERVENTIONS:
Biological: MGA271 — Up to 9 dose escalation cohorts will be enrolled to determine the maximum tolerated dose of MGA271. Patients with evidence of clinical benefit will be allowed to continue therapy at the same dose once per week for 3 weeks out of every 4-week cycle until documented progression.
  Patients treated in the Expansion Segment at the maximum administered dose will receive weekly, uninterrupted infusions of MGA271 in 8 week cycles for up to 12 cycles.

SUMMARY:
The purpose of this study is to evaluate the safety of MGA271 when given by intravenous (IV) infusion to patients with refractory cancer. The study will also evaluate how long MGA271 stays in the blood and how long it takes for it to leave the body, what is the highest dose that can safely be given, and whether it may have an effect on tumors.

DETAILED DESCRIPTION:
An open-label, multi-dose, single-arm, multi-center, Phase 1, dose-escalation study will be conducted to define the toxicity profile, maximum tolerated dose (MTD), pharmacokinetics (PK), immunogenicity, and potential antitumor activity of MGA271 in patients with refractory cancer that expresses B7-H3.

In the initial segments of the study, patients will be monitored for a minimum of four weeks after administration of the final dose of MGA271. Study assessments will include adverse event (AE) monitoring, electrocardiogram (ECG) monitoring, PK analysis of serum MGA271, determination of the serum concentration of soluble MGA271 and tumor markers, and an assessment of potential anti-MGA271 antibody [human anti-human antibody (HAHA)] response.

Tumor response assessments using Study Day 43 CT scans or MRI will be performed approximately six weeks after the first MGA271 dose for each patient. Patients with evidence of clinical benefit (partial or complete response or stable disease by RECIST or RANO Response criteria) will be allowed to continue therapy at the same dose, or at a reduced dose if warranted by dose limiting toxicity (DLT) or significant AE in Cycle 1. Subsequent cycles which will begin on Study Day 50 will consist of MGA271 administration on Study Days 1, 8, and 15 of each 28-day cycle, with tumor evaluation every other cycle. Responding patients may receive continued antibody therapy until evidence of progression of disease is documented or the patient experiences DLT.

In the Expansion Segment of the study, patients will receive weekly, uninterrupted infusions with an initial response assessment at 8 weeks. Tumor evaluation will be carried out by both RECIST and immune-related response criteria (irRC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed carcinoma (prostate cancer, renal cell carcinoma, head and neck cancer, triple-negative breast cancer, bladder cancer, non-small cell lung cancer) or melanoma that overexpresses B7-H3.
* Progressive disease during or after last treatment regimen.
* Appropriate treatment history for histological entity.
* ECOG Performance Status <= 1.
* Life expectancy >= 3 months.
* Measurable disease or evaluable disease with relevant tumor marker elevation.
* Acceptable laboratory parameters and adequate organ reserve.

Exclusion Criteria:

* Major surgery or trauma within four weeks before enrollment.
* Known hypersensitivity to murine or recombinant proteins, polysorbate 80, or any excipient contained in the drug formulation.
* Grade 3 colitis, hepatitis, pneumonitis uveitis, myocarditis, myositis, CNS toxicity or autoimmune related neuromuscular toxicity such as myasthenia gravis associated with the administration of an immune checkpoint inhibitor
* Second primary malignancy that has not been in remission for greater than 3 years. Treated non-melanoma skin cancer, cervical carcinoma in situ on biopsy, or squamous intraepithelial lesion on PAP smear, localized prostate cancer (Gleason score < 6), or resected melanoma in situ are exceptions and do not require a 3 year remission.
* Active viral, bacterial, or systemic fungal infection requiring parenteral treatment within four weeks of enrollment. Patients requiring any oral antiviral, fungal, or bacterial therapy must have completed treatment within one week of enrollment.
* Vaccination within 2 weeks of enrollment (except for annual flu vaccine).
* History of chronic or recurrent infections that require continual use of antiviral, antifungal, or antibacterial agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2011-07; Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Safety | Study Day 50 or 28 days after last infusion
  Adverse events, serious adverse events, ECG monitoring, adrenal function monitoring, monitoring for development of anti-drug antibodies

SECONDARY OUTCOMES:
Maximum tolerated dose | Study Day 50 or 28 days after last infusion

OTHER OUTCOMES:
Tumor response | Every 8 weeks
  Efficacy will be assessed every 8 weeks in the Expansion Segment according to immune-related response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — MacroGenics
Locations (12):
- United States (12):
  - UCLA Hematology-Oncology Clinic, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Chicago, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Neely Center for Clinical Cancer Research, Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Carolina Biooncology Institute, Huntersville, North Carolina
  - Hospital of the University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No